CLINICAL TRIAL: NCT04874324
Title: Phase-I Double-blind, Randomized, Placebo-controlled Single Center Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of Oral WCK 2349 Under Fasting Conditions in Adult Healthy Human Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of Oral WCK 2349
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: WCK 2349/ P-I/ MD/ 08
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — levonadifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WCK 2349 (Experimental): WCK 2349 800mg, 1000mg, and 1200mg . 1 dose given orally twice daily at 12 hourly interval for five days.
  Dosage form : Oral
  Interventions: Drug: WCK 2349 Oral
- Placebo (Placebo Comparator): Matching Placebo administered as Oral
  Interventions: Other: Placebo Oral

INTERVENTIONS:
Drug: WCK 2349 Oral — 1 dose given orally twice daily at 12 hourly interval for five days.
  Arms: WCK 2349
Other: Placebo Oral — Subjects will receive matching placebo
  Arms: Placebo

SUMMARY:
The present study is planned to assess the safety, tolerability and pharmacokinetic profile of WCK 2349 in US subjects with selected ascending multiple doses of WCK 2349 and to compare the safety, tolerability and pharmacokinetic data with the data observed in similar studies conducted in India.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy males or non-pregnant females
* Have a Body Mass Index (BMI) between 18 and 32 (both inclusive), calculated as weight in kg / height in m2
* Have no significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations and ECG recordings.
* Should test negative for drugs of abuse and urine alcohol test.

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to quinolones or any other related drugs.
* Any history or evidence of disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-03-17 (Actual); Primary Completion 2011-05-04 (Actual); Study Completion 2011-06-25 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety & tolerability of multiple doses of WCK 2349 | 12 days
  By monitoring the adverse events reported
To evaluate the pharmacokinetics of multiple doses of WCK 2349 | 5 days
  Measuring Cmax Maximum observed plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Ashima Bhatia, MD, Study Director — Wockhardt Ltd